CLINICAL TRIAL: NCT03065894
Title: Does Risk Stratification in Primary Care Combined With Stratified-specific Physical Therapy Care Improve Clinical Outcomes for Patients With Nonspecific Low Back Pain Compared to Those Who Receive Only Current Care?
Brief Title: Risk Stratification in Primary Care Combined With Stratified-specific Physical Therapy Care for Low Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of subject enrollment
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Sharon Henry, Therapy Research Educator, University of Vermont Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-494
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Low Back Pain
Keywords: stratified care; psychologically informed practice; matched care
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Prospective, longitudinal, pragmatic, non-randomized clustered, non-blinded, controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stratified Care (Experimental): In three "Participating Sites" from Family Medicine sites, the Keele STarT Back Screening Tool will be administered to patients with acute and chronic low back pain and based on patients' responses, patients will be stratified into one of three risk groups: low, medium or high-risk. Patients in the medium- and high-risk groups will be referred to physical therapy for a matched physical therapy (PT) intervention based on the risk strata. Patients in the low-risk group will be managed in Family Medicine with an intervention that includes advice, reassurance, patient education, and NSAIDs (with no referral for imaging or specialist care).
  Interventions: Other: Matched Physical Therapy Intervention
- Current Care (Active Comparator): In three "Comparator Sites" from Family Medicine, providers will give the current care at The University of Vermont Medical Center for patients with acute and chronic low back pain.
  Interventions: Other: Current Care in Family Medicine

INTERVENTIONS:
Other: Matched Physical Therapy Intervention — Patients who are medium-risk will receive up to 6-8 physical therapy (PT) visits over a 3 month period that is guided by published evidence based practice guidelines. The PT treatment will be tailored to the physical findings and specific patient needs, and appropriate exercises, spinal mobilization/manipulation, strengthening/stretching as well as a home program will be given to improve patient pain and function and reduce disability.
  Patients who are high-risk will receive the evidence based PT treatment as deemed necessary. In addition, the PT treatment will incorporate principles of psychologically informed practice to address psychosocial barriers (e.g., fear avoidance, anxiety, etc) that may be impeding disability reduction. This may include instruction on chronic pain rehabilitation techniques such as the use of: pacing in order to maintain or increase activity; graded activity principles in order to increase function; and pain education and understanding responses to pain.
  Arms: Stratified Care
Other: Current Care in Family Medicine — Patient education, medication management
  Arms: Current Care

SUMMARY:
This study aims to examine patient outcomes following risk stratification for low back pain in Family Medicine combined with either matched physical therapy (PT - i.e., stratified-specific PT) treatments or current treatment in primary care across The University of Vermont Health Network.

DETAILED DESCRIPTION:
The University of Vermont Health Network is a five hospital network that serves primarily a rural population of approximately 1 million people in Vermont and upstate New York. The primary aim of this prospective, longitudinal, pragmatic, non-randomized clustered, non-blinded, controlled trial is to examine whether PT treatment stratified to match the patient's risk factors based on the STarT Back Tool is more effective than the current treatment in primary care for non-specific low back pain (LBP) in improving short- (6 months) and long-term (12-month) patient outcomes (disability).

To do the risk stratification, investigators will use the STarT Back Tool which is designed for primary care settings and is validated for non-specific LBP (acute flare-ups or chronic pain). The tool is designed to identify the prognostic risk (low, medium, high) for progression to chronic LBP. In addition, the tool assists clinicians in decision making to ensure that low risk patients are not over treated or medicalized, that 'at risk' patients get access to the right provider early on and that enhanced care is given for complex cases. Thus, the tool assists in matching the 'right patient to the right treatment' at the 'right time' which is critical given the high prevalence and cost of LBP.

Patients with a primary diagnosis of LBP (acute flare-up or chronic) who are seen in any of the six Family Medicine sites will complete the STarT Back Tool and the Modified Low Back Pain Disability Questionnaire (mODI). With the non-randomized, cluster design, three of the Family Medicine sites are identified as "Participating Sites" and three are identified as "Comparator Sites." Patients with low back pain from "Participating Sites" who are stratified as medium- or high-risk patients will be referred to physical therapy (PT) for a matched (i.e., stratified-specific treatment). Those patients who are identified as low-risk will be retained in Family Medicine for management using advice, reassurance, patient education, NSAIDs (no imaging or specialist referral is encouraged). Patients with low back pain from "Comparator Sites" will be managed according to current care practices in Family Medicine. Using the mODI, the investigators will compare the two study arms at short- (6 months) and long-term points (12 months).

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of acute, chronic or non-specific LBP,
2. between 21 - 60 years of age,
3. able to stand and walk without assistance,
4. able to understand and read English,
5. able to understand and sign a consent form.

Exclusion Criteria:

1. active serious spinal complications such as tumor or infection,
2. active treatment for metastatic or bone cancer of the spine,
3. pregnancy or less than 6 months post-partum or less than 6 months post weaning.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Modified Low Back Pain Disability Questionnaire | 6 months
  Low back pain disability measure

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M Henry, PT, PhD, Principal Investigator — The University of Vermont Medical Center
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No